CLINICAL TRIAL: NCT06334094
Title: Assessing the Cognitive Benefits of Ozanimod and Their Brain-Biomarkers in MS
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The funding for the study was revoked. As such, the study is no longer being conducted.
Sponsor: The University of Texas at Dallas (Other)
Collaborators: Texas Institute for Neurological Disorders (Unknown)
Responsible Party: Principal Investigator, Dr. Bart Rypma, Professor, The University of Texas at Dallas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-23-486; IM047-1054 (Other Grant/Funding Number: Bristol Myers Squibb)
Record Dates: First submitted 2024-02-26; First posted 2024-03-27 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Multiple Sclerosis
Keywords: Zeposia; Ozanimod
MeSH Terms: conditions — Multiple Sclerosis | interventions — ozanimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ozanimod (Experimental): Participants will receive Ozanimod and work up to .92 mg. They will then take one pill daily for a duration of 12 months.
  Interventions: Drug: Ozanimod

INTERVENTIONS:
Drug: Ozanimod — A hard capsule that is taken daily for one year.
  Other Names: Zeposia

SUMMARY:
The primary objective of this study is to investigate the cognitive benefits of ozanimod in individuals with Multiple Sclerosis (MS). The study aims to understand the neural basis of cognitive improvement in Relapsing-Remitting MS patients under ozanimod treatment using neuroimaging and behavioral techniques to characterize the brain and behavioral changes due to ozanimod treatment.

DETAILED DESCRIPTION:
To assess MS patients' cognitive improvement while on ozanimod, the investigators will compare MS patients' baseline performance to the patients' performance following treatment on memory, processing speed, verbal ability and executive function. The investigators predict that cognitive performance will improve during the ozanimod treatment compared to the baseline. Baseline-treatment differences will be assessed using repeated-measures analysis of covariance (ANCOVA) while also controlling for effects of age, education, disease duration, and expanded disability status score (EDSS). The investigators predict that improved cognitive performance will be accompanied by improvements in brain structure (e.g., increased whole brain volume) and function metrics.

Thus, each MS patients' brain volume, white matter connectivity, lesion load, and resting BOLD at baseline, during treatment, and after ozanimod treatment will be measured. For each structure and function MR metric, baseline-treatment differences will be assessed using repeated-measures ANCOVA while also controlling for effects of age, education, disease duration, EDSS and brain parenchymal fraction (the ratio of functional brain tissue to whole brain volume).

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking Relapsing-Remitting MS (RRMS; intermittent symptom exacerbations followed by periods of remission) patients.
2. Male and female, between the ages of 18-55 years old will be recruited from the Texas Institute for Neurological Disorders (TIND) and MS Clinic of The University of Texas Southwestern. Study referrals will come from board-certified neurologists.
3. Patients will have a McDonald-criteria diagnosis of RRMS, be >30 days past exacerbation and corticosteroid treatment.
4. Included patients will also be free of substance abuse and significant medical, other neurological, or psychiatric conditions unrelated to their MS disease course.
5. Patient selection will be limited to patients that are treatment naïve (i.e., have not been previously treated for their MS) or require a change in treatment course.
6. A clinical determination is needed as to whether ozanimod is the best treatment for a patient or whether a patient requires treatment change to ozanimod.
7. All included participants will be right-handed and at least high-school educated.
8. Only patients who score above 25 on the Telephone Interview for Cognitive Status (TICS) will be included.

Exclusion Criteria:

1. During calibrated functional magnetic resonance imaging (fMRI) scanning, participants will inhale a carbon dioxide/room air solution to allow for calibration of BOLD signal. Thus, to ensure participant safety, the investigators exclude: smokers and those with MR-contraindicators, any participants with a history of respiratory or pulmonary problems (e.g., asthma, Chronic Obstructive Pulmonary Disease (COPD), sarcoidosis, tuberculosis), any participant with a history of cerebral vascular disease (e.g., cardiac disease, transient ischemic attack, migraines, stroke, arteriovenous malformation), any participant with a history of respiratory or pulmonary problems (e.g., asthma, Chronic Obstructive Pulmonary Disease (COPD), sarcoidosis, tuberculosis), and any participant with a history of cerebral vascular disease (e.g., cardiac disease, transient ischemic attack, migraines, stroke, arteriovenous malformation).
2. Participants that present with EKG abnormalities consistent with FDA labeling contained within the ozanimod guidelines will be excluded as these abnormalities may be indication of dangerous negative side effects upon ozanimod consumption. EKG abnormalities include presence of atrioventricular (AV) block, sick sinus syndrome, or sino-atrial block. Any experiences of myocardial infarction, unstable angina, stroke, transient ischemic attack, decompensated heart failure requiring hospitalization, or Class III or IV heart failure within the last 6 months will exclude the patient. Contraindicators of ozanimod that may be found in the blood sample include presence of varicella titers and enzyme/protein levels that indicate liver dysfunction. Thus, these participants will be excluded.
3. Patients who exhibit diseases other than MS that may be responsible for the patient's clinical, or MRI presentation will be excluded.
4. Patients who exhibit a history of hypersensitivity to ozanimod or any drugs of similar chemical classes (i.e., sphingosine phosphates) will be excluded.
5. Female participants who are pregnant or nursing will be excluded from the study. After the participant consents to being in the study, there will be a screening appointment to determine their eligibility, at which a pregnancy test will be provided. Other examinations, such as neurological assessments and EKGs, will occur at this appointment.
6. Patients who are not native-English speakers will be excluded, as their English ability may limit their understanding of the instructions and performance on the neuropsychological tests.
7. Patients who score below 25 on the Telephone Interview for Cognitive Status (TICS) will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Processing Speed/Symbol-Digit Modality Test (SDMT) Performance | 1 year
  SDMT is a neuropsychological assessment of processing speed in MS. The SDMT consists of 9 symbols that correspond to a number. Participants have 90 seconds to complete as many symbol to number associations as they can. Scoring is based on how many they can complete correctly in the span of 90 seconds. Therefore, to assess MS patients' cognitive changes while on ozanimod, MS patients' baseline performance to their performance following treatment on processing speed will be compared. The primary endpoint for this study will be a change from baseline in written SDMT performance of at least 4 points.

SECONDARY OUTCOMES:
Change in Volumetric Blood-Oxygen-Level-Dependent (BOLD) signal as Measured by Dual Echo Functional Magnetic Resonance Imaging (fMRI) | 1 year
  To assess the mechanisms by which ozanimod changes processing speed in MS, fMRI measures will be obtained, including the patients' volumetric BOLD signal. To assess metrics of MS patients' structural and functional changes while on ozanimod, MS patients' resting BOLD will be measured. In the context of the within-subjects design, comparisons will be performed between each of the MS patients to themselves by comparing their baseline and treatment-assessment MR metrics. Each MS patients' resting BOLD signal will be measured at baseline, during treatment, and after ozanimod treatment. Additionally, BOLD signal of ozanimod-responders to non-responders will be compared.
Change in Cerebral Blood Flow (CBF) as Measured by Dual Echo Functional Magnetic Resonance Imaging (fMRI) | 1 year
  To assess metrics of MS patients' neurophysiology changes while on ozanimod compared to baseline, MS patients' CBF during the treatment phase will be assessed for comparison to baseline. In the context of the within-subjects design, comparisons will be performed between each of the MS patients to themselves by comparing their baseline and treatment-assessment MR metrics.
Change in Cerebral Metabolic Rate of Oxygen (CMRO2) as Measured by Dual Echo Functional Magnetic Resonance Imaging (fMRI) | 1 year
  To assess metrics of MS patients' neurophysiology changes while on ozanimod compared to baseline, MS patients' CMRO2 and CBF/CMRO2 ratio (i.e., NVC) will be assessed during the treatment phase for comparison to baseline. In the context of the within-subjects design, comparisons will be performed between each of the MS patients to themselves by comparing their baseline and treatment-assessment MR metrics.
Change in Whole Brain Volume as Measured By Structural Magnetic Resonance Imaging | 1 year
  To assess metrics of MS patients' structural and functional changes while on ozanimod, the investigators will measure MS patients' brain volume. In the context of the within-subjects design, comparisons will be performed between each of the MS patients to themselves by comparing their baseline and treatment-assessment MR metrics.
Differences in Diffusion parameters of ozanimod-responders to non-responders as Measured By a Diffusion Kurtosis Resonance Imaging (DKI) | 1 year
  To assess metrics of MS patients' neurophysiology changes while on ozanimod compared to baseline, MS patients' diffusion parameters of ozanimod-responders to non-responders will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Bart Rypma, PhD, Principal Investigator — The University of Texas at Dallas
Locations (1):
- Center for Brain Health, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with BMS researchers.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: After one year; in perpetuity.
Access Criteria: Bristol Myers Squibb (BMS) employment